CLINICAL TRIAL: NCT03433573
Title: Paediatric Use of the Abbott Sensor Based Glucose Monitoring System - an Accuracy Evaluation
Brief Title: Paediatric Use of the Abbott Sensor Based Glucose Monitoring System
Acronym: PUGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADC-UK-VAL-17032
Record Dates: First submitted 2018-02-09; First posted 2018-02-14 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Abbott Sensor Based Glucose Monitoring System
  Interventions: Device: Abbott Sensor Based Glucose Monitoring System

INTERVENTIONS:
Device: Abbott Sensor Based Glucose Monitoring System — Subjects will wear the Abbott Sensor Based Glucose Monitoring System and will be asked to perform 4 blood glucose tests per day (pre-meal and before bedtime). Subjects will be asked to scan the sensor when each blood glucose test is performed.

SUMMARY:
Accuracy evaluation of the Abbott Sensor Based Glucose Monitoring System when used by children with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-17 years (inclusive).
* Have type 1 or type 2 diabetes using insulin administered by injections or continuous subcutaneous insulin infusion (CSII).
* Currently testing blood glucose levels at least twice per day.
* Each participant has an identified Caregiver aged ≥18 years.
* In the investigator's opinion, technically capable of using device (participant and/or caregiver).

Exclusion Criteria:

* Concomitant disease or condition that may compromise patient safety including and not limited to; cystic fibrosis, severe mental illness, known or suspected eating disorder or any uncontrolled long term medical condition.
* Currently prescribed oral steroid therapy for any acute or chronic condition.
* Currently receiving dialysis treatment or planning to receive dialysis during the study.
* Female participant known to be pregnant.
* Participating in another study of a glucose monitoring device or drug that could affect glucose measurements or management.
* Currently using a real-time or professional use continuous glucose monitoring (CGM) or FreeStyle Libre device or is planning to use one during the study, and unwilling to stop use of the device during the study.
* Known (or suspected) allergy to medical grade adhesives.
* In the investigator's opinion the participant or caregiver is unsuitable to participate due to any other cause/reason (both patient and caregiver considered).

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Point Accuracy Determined as % within Consensus Error Grid Zone A | Up to 35 days
  Point accuracy of Sensor based glucose values compared to capillary fingerstick blood glucose, determined as % within Consensus Error Grid Zone A.

CONTACTS AND LOCATIONS:
Locations (11):
- United Kingdom (11):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Pennine Acute Hospitals NHS Trust, Manchester
  - Northampton General Hospitals NHS Trust, Northampton
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Salisbury NHS Foundation Trust, Salisbury
  - Southampton University Hospitals NHS Trust, Southampton
  - Great Western Hospitals NHS Foundation Trust, Swindon
  - Taunton and Somerset NHS Foundation Trust, Taunton
  - St George's Healthcare NHS Trust, Tooting
  - Royal Cornwall Hospitals NHS Trust, Truro

IPD SHARING:
Plan to Share IPD: No